CLINICAL TRIAL: NCT05744752
Title: Protective Effects of Allium Sativum and Moringa Oleifera Extract in Alleviating Lead Induced Defects on Dental Enamel of Rabbits
Brief Title: Effects of Allium Sativum and Moringa Oleifera Extract on Dental Enamel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arslan Saleem (Other)
Collaborators: Baqai Medical University (Other)
Responsible Party: Sponsor-Investigator, Arslan Saleem, Statistical Officer, Rashid Latif Medical College
Organization: Rashid Latif Medical College (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Trial2022001
Record Dates: First submitted 2022-10-17; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Lead Poisoning
Keywords: Moringa oleifera extract; Allium sativum extract; Dental Enamel; Rabbits
MeSH Terms: conditions — Lead Poisoning | interventions — lead acetate

STUDY DESIGN:
Intervention Model Description: A total of 90 male rabbits of average weight 1-2 kg will be obtained from the animal house of COMSATS University, Lahore. These rabbits will be segregated into 06 groups, each group consisting of 15 rabbits. All rabbits will be kept safe in iron cages under controlled temperature (25±2 C), humidity (55 ± 5%), and 12-hour dark-light cycle. One week after their acclimatization into a new environment the trial will begin. All experimental protocols will be performed following the guidelines for the human use of laboratory animals established at COMSATS University, Lahore.
Who Masked: Participant, Outcomes Assessor
Masking Description: It is an animal model study and the investigator will mask the groups as "A, B, C, D, E, F" so the outcome assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Other): Control; Placebo 1ml NaCl 0.9% daily for 12 weeks
  Interventions: Other: Placebo
- Group B (Active Comparator): Pb Group; Lead acetate 19.5mg/kg b.w daily for 12 weeks
  Interventions: Other: Lead Acetate
- Group C (Experimental): Pb + Allium sativum extract; Lead acetate 19.5mg/kg b.w followed by Allium sativum(AS) extract 500 mg/kg b.w daily for 12 weeks
  Interventions: Other: Lead Acetate; Dietary Supplement: Allium sativum Extract
- Group D (Other): CPb + Moringa oleifera extract; Lead acetate 19.5mg/kg b.w followed by Moringa oleifera extract 400mg/kg b.w daily for 12 weeks
  Interventions: Other: Lead Acetate; Dietary Supplement: Moringa oleifera Extract
- Group E (Active Comparator): Allium sativum extract; Allium sativum extract 500mg/kg b.w daily for 12 weeks
  Interventions: Dietary Supplement: Allium sativum Extract
- Group F (Experimental): Moringa oleifera extract; Moringa oleifera extract 400mg/kg b.w daily for 12 weeks
  Interventions: Dietary Supplement: Moringa oleifera Extract

INTERVENTIONS:
Other: Lead Acetate — The oral LD50 of lead acetate is 390mg/kg body weight. The experimental group B, C, and D will receive a single dose of 19.5 mg/kg b.w (1/120th of LD50),31 daily dissolved in distilled water and given by oral gavage method for 12 weeks. Lead acetate Pb(CH3COO)2x3H2O, will be purchased from Sigma-Aldrich Chemie (Germany).
  Arms: Group B; Group C; Group D
Dietary Supplement: Moringa oleifera Extract — The method described by Hanaa Elgamily(32) with minor modifications. Fresh Leaves will be washed and dried in dry heat oven. All the preparation will be done in pharmacological department, University of Health Sciences in sterile environment. Dried leaves will be crushed to make fine powder. 1000 g powder of MO will be socked in 5000 ml of 70% ethanol (70% ethanol and 30% distilled water) for 72 hours at room temperature. Then mixture will be magnetically stirred for 24 hours and stored at 4oC for 48 hours to allow extraction of active ingredients. Then the mixture will be filtered twicely by using Whatman No 1 filter paper. The extract will be concentrated by rotary vacuum evaporator at 40 oC to evaporate the solvent. The extract will be freeze, dried and stored at -70 oC for use. Dose of MO extract will be 400 mg per kg.(33) body weight given daily in 1ml of distilled water by oral gavage method for 12 weeks.
  Arms: Group D; Group F
Dietary Supplement: Allium sativum Extract — Fresh Allium sativum bulbs will be selected for study. The cloves will be peeled, washed with distilled water and dried under shed. Then it will be chopped into small pieces. 1000g of chopped garlic will be crushed by mortar and passel. The garlic paste will be mixed with 5000 ml of 70% ethanol (70% ethanol and 30% distilled water) for 72 hours at room temperature. Rest the procedure is same as mentioned in moringa extract. Dose of 500 mg per kg(34) body weight garlic extract will be given daily in 1ml of distilled water.
  Arms: Group C; Group E
Other: Placebo — 1ml NaCl 0.9% daily for 12 weeks
  Arms: Group A

SUMMARY:
Primary objective is to observe the effects of lead on dental enamel of rabbit by measuring;

* Structural and morphological change by SEM, AFM
* Elemental composition by SEM-EDX
* Molecular composition and hydroxyapatite crystal changes by Raman Spectroscopy
* Blood parameters by serum analysis Secondary objectives includes
* To compare the protective effects of Allium sativum and Moringa oleifera on dental enamel defects due to lead
* To determine the beneficial effects of AS and MO extract in remineralization of dental enamel.

DETAILED DESCRIPTION:
This Animal experimental study will be carried out in animal House, University of Health Sciences, Lahore (UHS) and COMSATS University, Lahore. For this study fifty four healthy male, white NewZeeland rabbits (9 to 10 weeks) will be taken for the study. Rabbits will be randomly divided into 6 groups. Sample size will be 9 rabbits in each group. Experimental animals will be assigned number 1,2,3,4, till 54 using the random number generator and the randomly divided into six groups (n=9) and will be assigned as group A, B, C, D, E, and F. Healthy male, white New Zeeland rabbits weighing 1000-1200 grams (Age 9-10 weeks) will be selected from University of Veterinary and Animal Sciences, Lahore. The animals will be shifted to animal house of UHS. Animals will be kept in experimental research laboratory at controlled room temperature (22-24°C) and humidity (45-65 %) under 12/12 hours natural light and dark cycle for 2 weeks to acclimatize in new environment. All experimental animals will be fed on vegetables, fruits and distilled water ad libitum. At the end of 12 weeks, all the animals will be sacrificed under deep anesthesia. Ketamine hydrochloride 45 mg/kg b.w and xylazine 5 mg/kg b.w I/M will be given to maintain deep anesthesia. Afterwards, 20 mg xylazine was injected into the pinna vein to sacrifice the rabbits while they were anesthetized.(35).

Blood Sampling: The Central Auricular Artery(36) or lateral saphenous vein will be selected to collect 4 ml blood on day 0, after 8 weeks and at the end of 12 weeks. The sample will be collected in serum separating tube for investigations like blood lead count, alkaline phosphatase, calcium and phosphate level.

Tissue Sampling Technique:

A portion of 4x5 mm2 from middle third of crown labial surface will be taken for investigations. The cutting will be done by diamond disc and high speed turbine with irrigation of water to ovoid over heating of sample. Right mandibular incisors of all the rabbits will be selected for SEM and AFM. The left mandibular incisors of all the rabbits will be selected SEM-EDX and RMS analysis. All samples will be labeled and stored in sterilized container having 12% formalin for 72 hours.

Laboratory Processing:

1. Scan Electron Microscopy: Right mandibular incisor will be selected for SEM analysis. The structure and morphological features of enamel will be seen by its images. The sample will be washed with distilled water and will be dried by hot air blower at slow speed. Sixteen samples can be fixed on a sample stab at a time. Samples will be fixed on stab by double copper tape. The exposed stab will also be covered by copper tape and only the sample part will be left uncovered.

   Gold coating will be done in sputter coater machine to make the surface conductor for fine details of images. The sample stab will be place in sputter machine chamber and lid will be closed. Inside the chamber, vacuum will be created and argon gas will be filled. Potential of 40 volts will be given. By this plasma will be formed inside the chamber and the electrons of argon gas will strike on gold plate. The tiny gold particles will start sputtering on sample stab. Once gold coating will be done, the procedure will be reversed. The chamber will be filled with air and lid will be opened. Now the sample will be processed in NOVA NANOSEM 450 for ultrastructural details.
2. Energy Dispersive Spectroscopy: EDX will be used to study elemental composition of mineral contents. A detector of OXFORD X-ACT, PENTA FET will be attached with NOVA NANOSEM 450. The same sample used for SEM will also be used for SEM-EDX analysis. This will give details on the surface up to 2 micron thickness.
3. Atomic Force Microscope: AFM (SPM-9500J3, Shimadzu Corp, Japan) will be used for the assessment of morphological features of enamel surface. It provides the three-dimensional surface topography without any sample preparation. This microscopy is designed to scan the sample with a probe. Sample will be attached on stub, which will be fixed and manually adjusted. Laser adjustment will be done after determining probe frequency. Finally, scanning and image processing will be done with WinSPM system processing. For one representative sample, micrographs at six different areas (2.0×2.0 μm scan area) will be taken using AFM (SPM-9500J3, Shimadzu Corp, Japan) and AFM software (SPM-Offline, Shimadzu Corp, Japan).

   AFM creates 3D images of a surface by scanning a micron-size cantilever across the surface, which is typically made of silicon or silicon nitride, with a tip whose radius of curvature is ~10nm. The cantilever is deflected by the forces between the tip and the surface, which are ~nN and include contributions from electrostatic forces, solvation forces, Vander Waals interactions, and chemical bonding. This deflection of cantilever is measured by a laser spot reflecting from the top surface of the cantilever into an array of photodiodes, which provides images on the computer.
4. Raman spectroscopy: It is a non-destructive chemical analysis technique which provides detailed information about chemical structure, crystallinity and molecular interactions. The RMS will give us the details of the entire thickness of enamel about the molecular composition and its interaction of the sample. No special sample preparation will be needed for this analysis and the sample can also be used for other investigations. InVia Raman Microscope by RENISHAW UK will be used for this study. The laser intensity 488nm will be used for 10 seconds. The RMS will be done on 6 different spots and the average reading will be used in study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy rabbits
* Rabbits Age 9-10 weeks
* Weight 1000-1200 g will be selected

Exclusion Criteria:

* Diseased rabbit
* Age: More than 10 weeks and less than 9 weeks
* Weight more than 1200 g and less than 1000 g

Ages: 3 Months to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Healthy male rabbits of average weight 1-2 kg
Enrollment: 90 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Histological Outcomes | at the end of the study
  In this examination Odontoblastic zone, Cell nuclei Vacuolization of odontoblasts, Acute Inflammation, Chronic Inflammation, Apatite formation, Collagen crosslinking will be determined inform of normal or abnormal.

SECONDARY OUTCOMES:
Mineral Concentration | at the end of the study
  Mineral concentration like Ca/P etc. ratio will be assessed by SEM & EDX analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rashid Javaid, Ph.D scholar, Principal Investigator — Baqai Medical University
Locations (1):
- Baqai Medical University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data analysis will be presented in the form of graphs and tables in the thesis. The graphs will be generated from Energy-dispersive X-ray spectroscopy(EDX) and Scanning Electron Microscope (SEM) and will interpreted by the Expert.

REFERENCES:
- [Background] Du Toit N, Kempson SA, Dixon PM. Donkey dental anatomy. Part 2: Histological and scanning electron microscopic examinations. Vet J. 2008 Jun;176(3):345-53. doi: 10.1016/j.tvjl.2008.03.004. Epub 2008 Apr 18. PMID 18396075
- [Background] Six N, Lasfargues JJ, Goldberg M. Differential repair responses in the coronal and radicular areas of the exposed rat molar pulp induced by recombinant human bone morphogenetic protein 7 (osteogenic protein 1). Arch Oral Biol. 2002 Mar;47(3):177-87. doi: 10.1016/s0003-9969(01)00100-5. PMID 11839353
- [Result] Yu C, Abbott PV. An overview of the dental pulp: its functions and responses to injury. Aust Dent J. 2007 Mar;52(1 Suppl):S4-16. doi: 10.1111/j.1834-7819.2007.tb00525.x. PMID 17546858